CLINICAL TRIAL: NCT02044276
Title: A Randomized, Phase IIIB, Open-label, Two-arm, Multicenter, comparatiVe Study on Efficacy and Safety of Lipegfilgrastim (Lonquex, TEVA) in Comparison to Pegfilgrastim (Neulasta(R), Amgen) in Elderly Patients With Aggressive B Cell Non-HOdgkin Lymphomas at hIgh Risk for R-CHOP-21-inDuced Neutropenia - AVOID Neutropenia
Brief Title: A comparatiVe Study on Efficacy and Safety of Lipegfilgrastim in Comparison to Pegfilgrastim in Elderly Patients With Aggressive B Cell Non-HOdgkin Lymphomas at hIgh Risk for R-CHOP-21-inDuced Neutropenia
Acronym: AVOID
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XM22-ONC-305; 2013-001284-23 (EudraCT Number)
Record Dates: First submitted 2014-01-21; First posted 2014-01-23 (Estimated); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Aggressive B Cell Non-Hodgkin Lymphomas at High Risk for R-CHOP-21-induced Neutropenia
Keywords: Neutropenia; NHL; Non-Hodgkin lymphomas; R-CHOP-21
MeSH Terms: conditions — Neutropenia | interventions — pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lipegfilgrastim. (Experimental): subcutaneous (SC) injection of 6 mg lipegfilgrastim
  Interventions: Drug: lipegfilgrastim
- pegfilgrastim (Active Comparator): SC injection of 6 mg pegfilgrastim
  Interventions: Drug: pegfilgrastim

INTERVENTIONS:
Drug: lipegfilgrastim — 6 mg
  Other Names: XM22
  Arms: lipegfilgrastim.
Drug: pegfilgrastim — 6 mg
  Other Names: Neulasta®
  Arms: pegfilgrastim

SUMMARY:
The primary objective of the study is to demonstrate non-inferiority of lipegfilgrastim to pegfilgrastim for the duration of severe neutropenia in the first cycle of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated Independent Ethics Committee (IEC)-approved written informed consent
2. Age ≥65 years and ≤85 years
3. Histological documentation of aggressive B cell NHL
4. Planned to receive systemic anticancer therapy with at least 6 cycles of R-CHOP-21, according to local standards
5. ECOG score ≤2
6. Life expectancy of at least 3 months
7. Adequate bone marrow, renal and hepatic function within 14 days before start of chemotherapy
8. The patient is capable of understanding and complying with parameters as outlined in the protocol
9. Women of childbearing potential (not surgically sterile or 2 years postmenopausal) must use a medically accepted method of contraception and must agree to continue use of this method for the duration of the treatment and for 30 days after discontinuation of study drug.
10. The patient, if a man, is surgically sterile, or, if capable of producing offspring, is currently using an approved method of birth control and agrees to continued use of this method for the duration of the treatment (and for 90 days after taking the last dose of study

    * Other Criteria apply, please contact the investigator for more information

Exclusion Criteria:

1. Participation in a clinical study within 30 days before randomization
2. Any chemotherapy within the last 3 months before start of chemotherapy. A prephase to reduce tumor burden prior to start of R-CHOP is allowed.
3. The patient is a pregnant or lactating woman. (Any woman becoming pregnant during the study will be withdrawn from the study.)
4. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days before start of chemotherapy.
5. Active cardiac disease
6. Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within the 6 months before start of chemotherapy.
7. Ongoing infection, known history of human immunodeficiency virus (HIV) infection, tuberculosis, or chronic hepatitis B or C.
8. Patients with evidence or history of bleeding diathesis.
9. Non-healing wound, ulcer or bone fracture.
10. Renal failure requiring hemo- or peritoneal dialysis.
11. Any conditions that may interfere with the patient's participation in the study or evaluation of the study results.
12. Known hypersensitivity to any of the study drugs, study drug classes, or excipients in the formulation.
13. Any illness or medical conditions that are unstable or could jeopardize the safety of the patient and his/her compliance in the study.
14. Treatment with lithium at screening or planned during the study.

    * Other Criteria apply, please contact the investigator for more information

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 101 (Actual)
Dates: Start 2014-03-31 (Actual); Primary Completion 2017-08-29 (Actual); Study Completion 2018-04-24 (Actual)

PRIMARY OUTCOMES:
Duration of severe neutropenia (DSN) ANC <0.5 * 10^9/L | 3 weeks
  Grade 4 neutropenia measured in days

SECONDARY OUTCOMES:
Incidence of febrile neutropenia (FN) (strict definition) | 18 weeks
  Body temperature of >38.5°C for at least one hour and ANC<1*10^9/L
Incidence of FN | 18 weeks
  A single temperature of ≥38.3°C or ≥38.0°C for at least one hour and ANC <1 * 10^9/L
Incidence of very severe neutropenia | 3 weeks
  The occurrence of at least one incidence of ANC <0.1 * 10*9/L
Incidence of infections | 18 weeks
  Incidence and severity of infections
Time to ANC recovery | 3 weeks
  The time in days from start of chemotherapy administration until the ANC increases to ≥1.0 x 109/L, ≥1.5 x 109/L, and ≥2.0 x 109/L after the expected nadir
Summary of participants with adverse events | 9 Months

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (60):
- Germany (51):
  - Teva Investigational Site 32284, Aurich
  - Teva Investigational Site 32314, Bad Soden am Taunus
  - Teva Investigational Site 32267, Berlin
  - Teva Investigational Site 32277, Berlin
  - Teva Investigational Site 32292, Bochum
  - Teva Investigational Site 32400, Bonn
  - Teva Investigational Site 32318, Bonn
  - Teva Investigational Site 32294, Bottrop
  - Teva Investigational Site 32275, Cologne
  - Teva Investigational Site 32282, Dresden
  - Teva Investigational Site 32269, Dresden
  - Teva Investigational Site 32303, Dresden
  - Teva Investigational Site 32308, Frankfurt (Oder)
  - Teva Investigational Site 32302, Frankfurt-Hochst
  - Teva Investigational Site 32276, Frechen
  - Teva Investigational Site 32293, Freiburg im Breisgau
  - Teva Investigational Site 32290, Freiburg im Breisgau
  - Teva Investigational Site 32322, Fulda
  - Teva Investigational Site 32320, Fürth
  - Teva Investigational Site 32273, Goslar
  - Teva Investigational Site 32296, Gütersloh
  - Teva Investigational Site 32319, Halle
  - Teva Investigational Site 32272, Hamburg
  - Teva Investigational Site 32295, Heilbronn
  - Teva Investigational Site 32270, Herne
  - Teva Investigational Site 32401, Herne
  - Teva Investigational Site 32279, Hof
  - Teva Investigational Site 32297, Kaiserslautern
  - Teva Investigational Site 32310, Kassel
  - Teva Investigational Site 32280, Kiel
  - Teva Investigational Site 32309, Krefeld
  - Teva Investigational Site 32287, Lahr
  - Teva Investigational Site 32289, Langen
  - Teva Investigational Site 32313, Lebach
  - Teva Investigational Site 32311, Leer
  - Teva Investigational Site 32278, Leipzig
  - Teva Investigational Site 32281, Mülheim
  - Teva Investigational Site 32301, München
  - Teva Investigational Site 32274, Oldenburg
  - Teva Investigational Site 32306, Pößneck
  - Teva Investigational Site 32304, Ravensburg
  - Teva Investigational Site 32291, Rotenburg (Wümme)
  - Teva Investigational Site 32315, Singen
  - Teva Investigational Site 32300, Stade
  - Teva Investigational Site 32288, Stolberg
  - Teva Investigational Site 32268, Stuttgart
  - Teva Investigational Site 32321, Stuttgart
  - Teva Investigational Site 32305, Torgau
  - Teva Investigational Site 32266, Villingen-Schwenningen
  - Teva Investigational Site 32317, Villingen-Schwenningen
  - Teva Investigational Site 32286, Weiden
- Italy (4):
  - Teva Investigational Site 30061, Campobasso
  - Teva Investigational Site 30059, Milan
  - Teva Investigational Site 30063, Napoli
  - Teva Investigational Site 30062, Torino
- Spain (5):
  - Teva Investigational Site 31074, Barcelona
  - Teva Investigational Site 31071, Madrid
  - Teva Investigational Site 31070, Madrid
  - Teva Investigational Site 31073, Valencia
  - Teva Investigational Site 31072, Valencia

REFERENCES:
- [Derived] Link H, Illerhaus G, Martens UM, Salar A, Depenbusch R, Kohler A, Engelhardt M, Mahlmann S, Zaiss M, Lammerich A, Bias P, Buchner A. Efficacy and safety of lipegfilgrastim versus pegfilgrastim in elderly patients with aggressive B cell non-Hodgkin lymphoma (B-NHL): results of the randomized, open-label, non-inferiority AVOID neutropenia study. Support Care Cancer. 2021 May;29(5):2519-2527. doi: 10.1007/s00520-020-05711-7. Epub 2020 Sep 17. PMID 32944800